CLINICAL TRIAL: NCT03347760
Title: Monocentric Interventionnal Pilot Study Pilot Study Evaluating Somatostatin Receptor's PET Imaging to Detect Inflammatory Phases of Myocarditis
Brief Title: Pilot Study Evaluating Somatostatin Receptor's PET Imaging to Detect Inflammatory Phases of Myocarditis
Acronym: DOTAMIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Elodie CHEVALIER, Dr, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-002716-43
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Myocarditis
Keywords: 68-Ga-DOTATOC PET; Myocarditis
MeSH Terms: conditions — Myocarditis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): All included patients wil receive 68Ga-dotatoc-PET/CT suspected acute myocarditis in first and an other 68Ga-dotatoc-PET/CT 6 months later
  Interventions: Drug: DOTATOC-68Ga PET initial; Drug: DOTATOC-68Ga PET at 6 months; Biological: blood sample

INTERVENTIONS:
Drug: DOTATOC-68Ga PET initial — DOTATOC is a tracer of high affinity for the type 2 somatostatin receptors and is used for imaging of tumours which are expressing them, including endocrine tumours
  Other Names: Imaging PET/CT
Drug: DOTATOC-68Ga PET at 6 months — DOTATOC is a tracer of high affinity for the type 2 somatostatin receptors and is used for imaging of tumours which are expressing them, including endocrine tumours
  Other Names: Imaging PET/CT
Biological: blood sample — blood tests will be carried out during the control visit to ensure that biological parameters are normalized

SUMMARY:
Infectious myocarditis are frequent, most of the time viral and can evolve to cardiac insufficiency. The diagnosis is difficult because they can mime an acute coronary syndrome. Approximately 10 % of patients with acute infarction suspected, have a normal angiography, and half of them has in fact a myocarditis, as showed studies of cardiac MRI among which some realized in our department . However, anomalies observed in MRI are not specific and it is necessary to use multiple criterions. A new radiopharmaceutical, the 68Ga-DOTATOC, specific of somatostatin's receptors which are over expressed by the inflammatory cells, has recently showed the capacity to identify myocarditis, but only in a small group of 6 patients.

The investigators make assumptions:

1. this radiopharmaceutical is enough sensitive to detect most of the acute inflammatory myocarditis which are identified by the MRI and
2. it could maybe allow to identify myocarditis with a persistent subacute or chronic inflammation, which are difficult to identify with cardiac MRI, and it would be a new information able to guide the medical decision.

Primary objectif: to determine if PET with 68Ga-DOTATOC is enough sensitive to identify myocarditis in acute inflammatory phase by hospitalized patients with suspected acute infarction and with normal angiography and who have a high probability of myocarditis identified by MRI. Disease prevalence will be close to 100 % at baseline Secondary objectives: 1. Estimate the frequency of inflammatory forms (subacute or chronicle), with a 68Ga-DOTATOC PET at 3 to 5 months from baseline, when classic signs of acute inflammatory generally disappeared (CRP, Troponin-I, myocardial oedema in MRI).

2. Analyze the concordance of the results of 68Ga-DOTATOC TEP by two readers

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects who have given their written consent to participate in the study.
* Patients without history of heart disease, hospitalized for acute infarction suspected with positive troponine, normal or subnormal angiography and which have a high probability of acute inflammatory myocardities on the secondarily realized MRI (= 2 criteria of Lake Louise)
* No contraindication to perform a 68Ga-DOTATOC-PET .
* Patient belong to a social security scheme.

Exclusion Criteria:

* Patients under guardianship or curatorship.
* Pregnancy, breastfeeding and woman of childbearing age without effective contraception
* Impossibility to perform a PET with 68Ga-DOTATOC (patient agitated).
* Impossibility to schedule PET/CT before the deadline = in 7 days since the beginning of the hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Presence of a significant myocardial retention of 68Ga-DOTATOC during initial staging. Sensibility calculation | at baseline
  The criterion of positivity will be that of a visually detectable and quantitatively significant area of myocardial uptake, which will be defined by a measurement of the Standardized Uptake Value (SUV) at least 30% higher than that of the blood signal obtained at the center of the left ventricular cavity. This threshold was chosen based on measurements already published in a small pilot study.

SECONDARY OUTCOMES:
Frequency of a significant myocardial retention of 68Ga-DOTATOC during initial staging | 6 months
  a visually detectable and quantitatively significant area of myocardial uptake, which will be defined by a measurement of the Standardized Uptake Value (SUV) at least 30% higher than that of the blood signal obtained at the center of the left ventricular cavity. This threshold was chosen based on measurements already published in a small pilot study.
  a visually detectable and quantitatively significant area of myocardial uptake, which will be defined by a measurement of the Standardized Uptake Value (SUV) at least 30% higher than that of the blood signal obtained at the center of the left ventricular cavity. This threshold was chosen based on measurements already published in a small pilot study.
  visually detectable and quantitatively significant area of myocardial uptake, which will be defined by a measurement of the Standardized Uptake Value (SUV) at least 30% higher than that of the blood signal obtained at the center of the left ventricular cavity.

CONTACTS AND LOCATIONS:
Overall Officials: Elodie CHEVALIER, MD, Principal Investigator — CHRU de NANCY
Locations (1):
- Véronique ROCH, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Derived] Larive T, Boursier C, Claudin M, Varlot J, Filippetti L, Huttin O, Roch V, Imbert L, Doyen M, Fraix A, Mandry D, Chevalier E, Marie PY. Persistent somatostatin PET signs of inflammatory cells 4 to 5 months after acute myocarditis are linked to a poorer recovery of cardiac function. Eur J Nucl Med Mol Imaging. 2025 Jul;52(9):3395-3403. doi: 10.1007/s00259-025-07202-5. Epub 2025 Mar 22. PMID 40119896